CLINICAL TRIAL: NCT03976531
Title: Multidisciplinary Development of the Geriatric Core Dataset for Clinical Research in Older Patients With Cancer: A French Initiative With International Survey
Brief Title: Geriatric Core Dataset (G-CODE) for Clinical Research in Elderly Cancer Patients
Acronym: G-CODE
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Plate-forme PACAN (Elderly and Cancer Platform) (Other); European Georges Pompidou Hospital (Other); Hospital Ambroise Paré Paris (Other); Institut Curie (Other); Centre Leon Berard (Other); Institut Claudius Regaud (Other); Saint-Louis Hospital, Paris, France (Other); Hospital Avicenne (Other); Göteborg University (Other); Oslo University Hospital (Other); City of Hope Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: IB2017-GCODE
Record Dates: First submitted 2019-05-23; First posted 2019-06-06 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Cancer
Keywords: cancer; elderly; randomized trial; consensus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly cancer patients included in randomized controlled trials

SUMMARY:
Older adults with cancer remain underrepresented in cancer clinical trials that establish new standards of care. Geriatric assessment (GA) is defined by geriatricians as a multidimensional interdisciplinary assessment of the general health stat us of the older patient, reviewing the medical, psychosocial, functional and environmental domains. For each domain, several tools are available, but consensus is lacking on which tool to use and the optimal cut-offs or threshold scores. The literature supports the prognostic value of the GA and its utility in weighing the benefits and risks of cancer treatments in older adults. However, GA has not been implemented in routine oncology practice or in cancer clinical trials.

The objective of this project is to develop a set of geriatric data, the Geriatric Core Dataset (G-CODE), to be collected in cancer trials of older patients. The methods rely on a consensus process involving international experts in the field of oncology and geriatrics.

DETAILED DESCRIPTION:
Although cancer is prevalent in the older segment of the population, older adults with cancer remain underrepresented in cancer clinical trials that establish new standards of care. As a result, robust data on the benefit/risk balance are lacking for many treatment strategies in these patients.

Ageing is a heterogeneous process that stresses the clinical need to identify comorbid conditions and ageing-related physiologic changes, both well-known factors increasing the risk of treatment side-effects and poor outcomes.

Geriatric assessment (GA) is defined by geriatricians as a multidimensional interdisciplinary assessment of the general health stat us of the older patient, reviewing the medical, psychosocial, functional and environmental domains. For each domain, several tools are available, but consensus is lacking on which tool to use and the optimal cut-offs or threshold scores. The literature supports the prognostic value of the GA and its utility in weighing the benefits and risks of cancer treatments in older adults. However, GA has not been implemented in routine oncology practice or in cancer clinical trials.

In 2011, after a workshop on clinical trial methodology in older adults with cancer, the Elderly Task Force of the European Organization for Research and Treatment of Cancer (EORTC) recommended the use of a standardised minimum data set (minDS) for assessing the global health and functional status of older populations. This minDS consisted of the G8 screening tool, the Instrumental Activities of Daily Living Following a consensus approach, a panel of 14 geriatricians from oncology clinics identified seven domains of importance in geriatric assessment. Based on the international recommendations, geriatricians selected the mostly commonly used tools/items for geriatric assessment by domain. The Geriatric Core Dataset (G-CODE) was progressively developed according to RAND appropriateness ratings and feedback during three successive Delphi rounds. The face validity of the G-CODE was assessed with two large panels of health professionals (55 national and 42 international experts) involved both in clinical practice and cancer trials.

ELIGIBILITY:
* cancer specialists (medical oncologists, surgeons, radiation oncologists, geriatricians, disease-oriented oncologists, clinical oncologists)
* clinical research associates
* nurses.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The panel of experts (cancer specialists, clinical research associates, nurses) was in charge of assessing the the relevance and approppriateness of the selected tools to include in the Geriatric Core Data Set (G-Code).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-01-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Mathoulin-Pélissier, MD/PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Paillaud E, Soubeyran P, Caillet P, Cudennec T, Brain E, Terret C, Etchepare F, Mourey L, Aparicio T, Pamoukdjian F, Audisio RA, Rostoft S, Hurria A, Bellera C, Mathoulin-Pelissier S; G-CODE collaborators. Multidisciplinary development of the Geriatric Core Dataset for clinical research in older patients with cancer: A French initiative with international survey. Eur J Cancer. 2018 Nov;103:61-68. doi: 10.1016/j.ejca.2018.07.137. Epub 2018 Sep 11. PMID 30212804

RESULTS

PARTICIPANT FLOW:
Groups:
- National Panel of Experts: National panel of experts involved in the scoring of the items/tools to be included in the G-CODE.
Period: Overall Study
Arm/Group | National Panel of Experts
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Age, Customized [Count of Participants; unit: Participants]
  >= 18 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Experts Who Considered That the Question "Do You Live Alone ?" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

2. Primary Outcome: Number of Experts Who Considered That the Question "do You Have a Person or Caregiver Able to Provide Care and Support" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

3. Primary Outcome: Number of Experts Who Considered That the Tool "ADL (Activities of Daily Living)" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

4. Primary Outcome: Number of Experts Who Considered That the Tool "4-IADL (Instrumental Activities of Daily Living)" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

5. Primary Outcome: Number of Experts Who Considered That the Test "Timed Up and Go" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

6. Primary Outcome: Number of Experts Who Considered That the Items "Weight Loss During the Past 6 Months and Body Mass Index (BMI)" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

7. Primary Outcome: Number of Experts Who Considered That the Item "One Cognitive Scale (Mini-Cog)" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

8. Primary Outcome: Number of Experts Who Considered That the Item "Char Lson Comorbidity Index" Should be Retained in the G-CODE
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | National Panel of Experts
Number analyzed (Participants) | 42
Participants | 42

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | National Panel of Experts
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes